CLINICAL TRIAL: NCT02819739
Title: Impact of Hyperoxia During Cardiopulmonary Bypass in the Occurrence of Cardiovascular Complications After Cardiac Surgery
Brief Title: Impact of Hyperoxia During Cardiopulmonary
Acronym: CARDIOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2014_843_0006; 2014-001403-44 (EudraCT Number)
Record Dates: First submitted 2015-01-05; First posted 2016-06-30 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Cardiac Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- normoxia (Experimental): During cardiopulmonary bypass inspired fraction of oxygen is adapted to maintained a oxygen arterial pressure below 150 mmHg.
  Interventions: Drug: medical oxygen
- hyperoxia (Active Comparator): During cardiopulmonary bypass inspired fraction of oxygen is set to 100 %.
  Interventions: Drug: medical oxygen

INTERVENTIONS:
Drug: medical oxygen

SUMMARY:
The hypothesis implies that this work is the use of hyperoxia during cardiopulmonary bypass by his heart preconditioning effect is associated with a lower incidence of cardiac arrhythmias (atrial fibrillation, tachycardia or ventricular fibrillation) and lesions of myocardial ischemia-reperfusion injury in cardiac surgery postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Major patient ≥ 18 years
* Patient operated cardiac surgery for myocardial revascularization (CABG) or surgical correction of valvular or combined surgery (CABG and valve disease) or ascending aortic surgery
* Signed Consent
* Affiliation to social security

Exclusion Criteria:

* Permanent atrial fibrillation
* Cordarone therapy,
* Pregnant woman
* Patient under guardianship or trusteeship or private public law
* Internal pacemaker
* Hypothermia,
* Patient refusal,
* Cardiac surgery without extracorporal circulation (ECC),
* Participation in another study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Occurred within 15 days after surgery, disorders of heart rhythm (atrial fibrillation, tachycardia or ventricular fibrillation) | 15 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Osama ABOU ARAB, Doctor, Principal Investigator — CHU Amiens-Picardie
Locations (2):
- France (2):
  - CHU Amiens-Picardie, Amiens
  - CHU Dijon-Bourgogne, Dijon

REFERENCES:
- [Derived] Abou-Arab O, Huette P, Martineau L, Beauvalot C, Beyls C, Josse E, Touati G, Bouchot O, Bouhemad B, Diouf M, Lorne E, Guinot PG. Hyperoxia during cardiopulmonary bypass does not decrease cardiovascular complications following cardiac surgery: the CARDIOX randomized clinical trial. Intensive Care Med. 2019 Oct;45(10):1413-1421. doi: 10.1007/s00134-019-05761-4. Epub 2019 Oct 1. PMID 31576438